CLINICAL TRIAL: NCT02987010
Title: A Phase 2 Study of the IDH1 Inhibitor, IDH305, for the Treatment of IDH1 Mutated Low Grade Glioma Patients Who Have Measurable 2HG by MR Spectroscopy
Brief Title: Phase 2 Study of IDH305 in Low Grade Gliomas
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor did not want to move forward with protocol; study was never opened.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 102016-038
Record Dates: First submitted 2016-11-21; First posted 2016-12-08 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort A (Experimental): Neoadjuvant administration of IDH305 at 550 mg BID for 6 weeks followed by surgical resection at 6 weeks. If there is no evidence of progressive disease at 6 weeks (clinical, radiographic or histopathologic exam), the patient will continue on IDH305 at 550 mg BID post-operatively for a maximum of 11 additional 28 day cycles. Subsequent assessment of disease will occur every 2 months starting in Cycle 2.
  Interventions: Drug: IDH305
- Cohort B (Experimental): Patients who have inoperable tumors but measurable 2HG pre-treatment will be treated with IDH305 at 550 mg BID x 6 weeks. If there is adequate sustained knockdown of 2HG on MRS and disease is stable or improved, then the patient will continue on treatment for a maximum of 11 additional 28 day cycles.
  Interventions: Drug: IDH305

INTERVENTIONS:
Drug: IDH305 — Isocitrate Dehydrogenase 1 inhibitor

SUMMARY:
Cohort A - neoadjuvant administration of IDH305 at 550 mg BID for 6 weeks followed by surgical resection at 6 weeks. If there is no evidence of progressive disease at 6 weeks (clinical, radiographic or histopathologic exam), the patient will continue on IDH305 at 550 mg BID post-operatively for a maximum of 11 additional 28 day cycles. Subsequent assessment of disease will occur every 2 months starting in Cycle 2.

Cohort B - patients who have inoperable tumors but measurable 2HG pre-treatment will be treated with IDH305 at 550 mg BID x 6 weeks. If there is adequate sustained knockdown of 2HG on MRS and disease is stable or improved, then the patient will continue on treatment for a maximum of 11 additional 28 day cycles.

DETAILED DESCRIPTION:
IDH1 mutations are thought to be among the earliest mutations occurring during transformation of glial cells into gliomas and dependence on the IDH-2HG pathway for survival and growth may be most relevant during the indolent phase of low grade tumor growth. However, the preclinical workup of IDH inhibitors was technically unable to assess low grade gliomas because the cells do not grow in vitro and so cannot be cultured, and the cells have such a low proliferation rate that they do not grow in mouse in vivo models. Despite this, Dr. Maher and colleagues have studied low grade metabolism in low grade gliomas in vivo, in patients undergoing surgical resection and infused with 13C-glucose or 13C-acetate. 13C-labeled tumor can be studied by 13C-nuclear magnetic resonance (NMR) ex vivo. 13C-NMR data from IDH-mutated low grade gliomas demonstrate that these tumors are highly metabolically active, capable of oxidizing both glucose and acetate while these substrates also contribute carbon to actively making 2HG (manuscript in preparation). These data strongly suggest that the low grade tumors may be dependent on the IDH pathway for maintaining the altered metabolic state of the cell and altered epigenome necessary for tumor growth. Treating low grade gliomas during the period of indolent growth poses a challenge in terms of evaluating a molecular targeted therapy for response and survival. Standard MRI assessment for low grade gliomas based on T2/FLAIR signal can be difficult to quantitate and reflects additional non-specific changes in the tumor microenvironment including edema and reactive gliosis. This is exacerbated by the natural history of these tumors for which there may be no change in tumor size over years. Added to this is the uncertainty that a drug was able to penetrate the blood brain barrier, enter the tumor and inhibit the target. To date, there is no non-invasive way to determine target inhibition, leaving the patients on a drug that may not inhibit the target and the investigator unsure if data being obtained reflects true activity. The current clinical trial addresses these challenges through a neoadjuvant clinical trial that combines non-invasive evaluation of 2HG by MRS to assess target inhibition within 1 week of study entry and direct tumor tissue analysis after 6 weeks on study in the surgical cohort. The comprehensive planned tissue analysis is designed to assess the impact of IDH305 on metabolic pathways, the epigenome and transcriptome, in addition to standard assessment of cellular proliferation and cell kill. A second cohort of patients, the non-surgical cohort, will include patients with a presumptive diagnosis of IDH-mutated glioma based on elevated 2HG on screening 2HG MRS but without a surgical resection planned because of perceived high risk of the procedure. It is anticipated that ~ 93% of these patients will have an IDH1 mutation and thus treatment with the IDH1 selective inhibitor will knockdown 2HG. For patients with an IDH2 mutation (~7-8%), we anticipate that there will be no change in 2HG. These patients will come off study, sparing them any potential toxicity without potential benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to any screening procedures that are not part of standard of care.
2. Age greater than or equal to 18 years.
3. Male or female of any racial or ethnic origin.
4. Measurable 2HG by MR Spectroscopy (above threshold of 1mM, established at UTSW).
5. Karnofsky Performance Status > 70%.
6. Measurable disease per RANO criteria.
7. Female subjects with reproductive potential must have a negative serum pregnancy test within 7 days prior to start of therapy. Subjects with reproductive potential are defined as one who is biologically capable of becoming pregnant. Women of childbearing potential as well as fertile men and their partners must agree to abstain from sexual intercourse or to use two effective forms of contraception during the study and for 30 days (females and males) following the last dose of IDH305.

Exclusion Criteria:

1. 2HG by MR Spectroscopy below 1 mM.
2. Patients who are currently receiving treatment with a prohibited medication or herbal remedy that cannot be discontinued at least one week prior to the start of treatment.
3. Narrow therapeutic index substrates of CYP3A, CYP2C9, CYP2C19, and CYP2C8.
4. Medications, herbs and supplements that are strong inhibitors and strong inducers of CYP3A.
5. Other herbal preparations and supplements.
6. Inhibitors of UGT1A1.
7. Patients who have out of range laboratory values defined as:

   * Absolute neutrophil count (ANC) <1.0 x 109/L
   * Hemoglobin (Hgb) <8 g/dL
   * Platelets <75 x 109/L
   * Total bilirubin > ULN
   * AST or ALT >3 x ULN
   * Serum creatinine >1.5 x ULN
8. Karnofsky Performance Status < 70%.
9. Malignant disease other than that being treated in this study. Exceptions to this exclusion include the following: malignancies that were treated curatively and have not recurred within the prior 2 years; completely resected basal cell and squamous cell skin cancers; any malignancy considered to be indolent and that has never required therapy; and completely resected carcinoma in situ of any type.
10. Patients with corrected QT using the Fridericia correction (QTcF) > 470 msec, or other clinically significant, uncontrolled heart disease, including acute myocardial infarction or unstable angina < 3 months prior to the first dose of IDH305.
11. Any other medical condition that would, in the investigator's judgment, prevent the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures such as the presence of other clinically significant cardiac, respiratory, gastrointestinal, renal, hepatic or neurological disease.
12. Patients with Gilbert's syndrome or other heritable diseases of bile processing.
13. Patients who are claustrophobic or who have other contraindications to MRI, such as an implanted pacemaker device, vascular clips, prosthetic valves, or otologic implants.
14. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
15. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 30 days after the use of the investigational medication. Highly effective contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the patient). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment Male sterilization (at least 6 months prior to screening). The vasectomized male partner should be the sole partner for that patient.
    * Combination of any two of the following (a+b, a+c, or b+c):

      a. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal, for example hormone vaginal ring or transdermal hormone contraception.
    * In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

      b. Placement of an intrauterine device (IUD) or intrauterine system (IUS). c. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
16. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
17. Sexually active males must use a condom during intercourse while taking the drug and for 30 days after stopping treatment and should not father a child in this period. A condom is required to be used also by vasectomized men as well as during intercourse with a male partner in order to prevent delivery of the drug via semen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
IDH305 treatment of 2HG | Twice a day for 6 weeks for a maximum of 11 additional 28 day cycles
  Number of participants treated with IDH305 leads to sustained knockdown of 2HG by MR spectroscopy from Baseline.
2HG response to IDH305 | Every 112 days, up to 365 days
  Number of participants with radiographic and clinical response to knockdown of 2HG by IDH305 compared to Baseline.

IPD SHARING:
Plan to Share IPD: No